CLINICAL TRIAL: NCT07163559
Title: Effectiveness of Client-Centered Coping Skills Training in Migraine: A 6-Month Follow-Up, Double-Blind, Randomized Controlled Trial
Brief Title: Coping Skills for Migraine: A 6-Month Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Etkin Bagi, Msc Occupational Therapist, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HU-ERG-EB-03
Record Dates: First submitted 2025-09-01; First posted 2025-09-09 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Migraine
Keywords: Migraine; Coping skills; Quality of life; Pain; Disability; Randomized controlled trial
MeSH Terms: conditions — Migraine Disorders; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention group (Experimental): CST aims to improve physical/mental health in chronic headache patients by reducing pain intensity, migraine attacks, and medication use. The program includes 8 sessions (2/week) covering:
  Client-centered problem-solving & migraine education (COPM-based), Activity pacing, stress management, and healthy habits, Energy conservation techniques, Social participation, Program evaluation. Session durations: Session 1 (45 min), Sessions 2-6 (60-75 min), Sessions 7-8 (60 min).
  Interventions: Behavioral: coping skills training
- control group (No Intervention)

INTERVENTIONS:
Behavioral: coping skills training — CST aims to improve physical/mental health in chronic headache patients by reducing pain intensity, migraine attacks, and medication use. The program includes 8 sessions (2/week) covering:
  Client-centered problem-solving & migraine education (COPM-based), Activity pacing, stress management, and healthy habits, Energy conservation techniques, Social participation, Program evaluation. Session durations: Session 1 (45 min), Sessions 2-6 (60-75 min), Sessions 7-8 (60 min).
  Arms: intervention group

SUMMARY:
This study aimed to investigate the effects of client-centered coping skills training on pain, quality of life, disability level, and coping skills in individuals with migraine over a 6-month follow-up period.

DETAILED DESCRIPTION:
Migraine is a significant public health issue characterized by frequently unilateral, recurrent, throbbing headaches. International Headache Disorders define migraine as a headache lasting 4-72 hours, accompanied by nausea, vomiting, phonophobia, or photophobia. Recurrent attacks can make it difficult to perform routine daily activities and movements. The World Health Organization lists migraine as one of the most disabling diseases. Approaches to treating migraine include pharmacological and non-pharmacological interventions. Non-pharmacological approaches aim to increase an individual's coping skills using exercise, stress management, and cognitive-behavioral therapy, which involve physical, mental, and cognitive interventions. While these approaches are practical individually, due to the impact of migraine on an individual's entire life, combined and client-centered approaches are needed.

Coping skills training (CST) has been shown to improve the physical and mental health and well-being of individuals with chronic headaches, significantly reducing pain intensity, migraine attacks, and medication use. It also aims to help individuals adapt to life more productively. Despite its positive effects, limited studies examine the impact of CST on individuals' coping skills and quality of life. A person-centered approach that combines various intervention components can enhance personal control and effectiveness in managing headaches. Due to the unpredictable timing of severe migraine attacks and the variable frequency of symptoms, client-centered coping skills training is recommended for managing migraines. Therefore, this study aimed to investigate the effects of client-centered coping skills training on pain, quality of life, disability level, and coping skills in individuals with migraine over a 6-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of migraine based on the International Classification of Headache Disorders (ICHD-3 beta) criteria,
* age between 18 and 65 years,
* literacy

Exclusion Criteria:

* psychiatric disorders,
* traumatic brain injury,
* other types of headaches,
* use of antidepressants, analgesics, anti-inflammatory drugs, or abusive substances (1 week before and during the treatments),
* any additional treatment for migraine during the study period,
* breastfeeding,
* pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | six months
  Visual Analog Scale (VAS) is a pain intensity measurement scale. It consists of a horizontal line 10 cm in length. The participants were asked to indicate their average pain over the last month by drawing a line, placing a dot, or marking a point on this line. The value of 10 on the line's right side represents severe pain, while the value of 0 on the left side represents the absence of pain. This indicates that the maximum degree of pain is at the far right boundary, and the minimum is at the far left boundary. The length of the distance between the point the participants mark on the line and the point representing the absence of pain indicates the intensity of their pain. The internal consistency of the VAS scale has been found to be 0.82 .

SECONDARY OUTCOMES:
Nottingham Health Profile (NHP) | six months
  Nottingham Health Profile (NHP) is a quality of life scale used to measure individuals' perceived health problems and how they affect their daily activities. It was developed by a group of researchers in the Department of Community Health at the University of Nottingham, England, in 1975 and completed in 1981. The NHP includes 38 items under six main headings of health: pain (8 items), emotional reactions (9 items), sleep (5 items), social isolation (5 items), physical mobility (8 items), and energy level (3 items). Individuals respond with either a yes or no to the item that is appropriate for them. Scores for each parameter range from 0 to 100, with a maximum total score of 600. The higher the score for any parameter, the more severe the perceived problem. This study used the Turkish version of the NHP, which has demonstrated excellent internal consistency with a Cronbach's alpha of 0.82.
Migraine Disability Assessment Scale (MIDAS) | six months
  The Migraine Disability Assessment Scale (MIDAS) is used to evaluate disability caused by migraine. It is a valid and reliable scale developed by Stewart et al. to investigate the impact of migraine over the past three months. MIDAS's 1st, 3rd, and fifth questions provide the number of days missed due to migraine-related absence from school/work, household, and leisure activities. The 2nd and 4th questions provide the number of days with a 50% reduction in work/school performance due to migraine. This study used the Turkish version of MIDAS, which demonstrated good test-retest reliability with a value of 0.77.
Coping Orientation to Problems Experienced Inventory (Brief-COPE) | six months
  Coping Orientation to Problems Experienced Inventory (Brief-COPE) assesses individuals' coping styles. It consists of 14 subscales, each containing two items, for a total of 28 items, to evaluate active coping, planning, using instrumental support, using emotional support, venting, self-distraction, behavioral disengagement, self-blame, positive reframing, humor, substance use, denial, acceptance, and religion coping. Each subscale is evaluated separately. The scale items include 4-point Likert-type response options, with responses ranging from "4. Mostly true" to "1. Not at all true." Low scores indicate less use of the coping style, while high scores indicate greater use. This study used the Turkish version of the Brief COPE, which demonstrates a high internal consistency with a Cronbach alpha value of 0.85.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No